CLINICAL TRIAL: NCT01965210
Title: The Combined Effect of Dietary Fibre and Plant Protein on Appetite and Metabolic Function After Short-Term Consumption
Brief Title: The Effect of Dietary Fibre and Plant Protein on Appetite and Metabolic Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swedish University of Agricultural Sciences (Other)
Collaborators: Uppsala University (Other)
Responsible Party: Principal Investigator, Isabella Lee, PhD student, Swedish University of Agricultural Sciences
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: SLU-IL-S1
Record Dates: First submitted 2013-09-16; First posted 2013-10-18 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-10

CONDITIONS: Appetite Regulation
Keywords: Rye; Fermentable dietary fibre; Inulin; Plant protein; Gluten; Porridge; Bread; Appetite; Satiety; Hunger; Desire to eat; Metabolism; Glucose; Insulin; Gut hormones; Metabolomics; Gastric emptying rate; Breath hydrogen and methane excretion
MeSH Terms: conditions — Insulin Resistance | interventions — Inulin; Glutens

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- Rye + high dose inulin + low dose gluten (Experimental): Rye porridge supplemented with a high dose of the fermentable dietary fibre inulin and low dose of the plant protein gluten.
  Interventions: Other: Rye + equal doses of inulin & gluten; Other: Rye + low dose inulin + high dose gluten; Other: Large non-supplemented rye; Other: Small non-supplemented rye; Other: Refined wheat bread
- Rye + equal doses of inulin & gluten (Experimental): Rye porridge supplemented with equal doses of the fermentable dietary fibre inulin and the plant protein gluten.
  Interventions: Other: Rye + high dose inulin + low dose gluten; Other: Rye + low dose inulin + high dose gluten; Other: Large non-supplemented rye; Other: Small non-supplemented rye; Other: Refined wheat bread
- Rye + low dose inulin + high dose gluten (Experimental): Rye porridge supplemented with a low dose of the fermentable dietary fibre inulin and a high dose of the plant protein gluten.
  Interventions: Other: Rye + high dose inulin + low dose gluten; Other: Rye + equal doses of inulin & gluten; Other: Large non-supplemented rye; Other: Small non-supplemented rye; Other: Refined wheat bread
- Large non-supplemented rye (Experimental): Large portion of rye porridge without supplements.
  Interventions: Other: Rye + high dose inulin + low dose gluten; Other: Rye + equal doses of inulin & gluten; Other: Rye + low dose inulin + high dose gluten; Other: Small non-supplemented rye; Other: Refined wheat bread
- Small non-supplemented rye (Experimental): Small portion of rye porridge without supplements.
  Interventions: Other: Rye + high dose inulin + low dose gluten; Other: Rye + equal doses of inulin & gluten; Other: Rye + low dose inulin + high dose gluten; Other: Large non-supplemented rye; Other: Refined wheat bread
- Refined wheat bread (Active Comparator): Refined wheat bread.
  Interventions: Other: Rye + high dose inulin + low dose gluten; Other: Rye + equal doses of inulin & gluten; Other: Rye + low dose inulin + high dose gluten; Other: Large non-supplemented rye; Other: Small non-supplemented rye

INTERVENTIONS:
Other: Rye + high dose inulin + low dose gluten — In a randomized cross-over design each subject receive one of six iso-caloric breakfasts on six different occasions, separated by 1 w wash-out.
  Arms: Large non-supplemented rye; Refined wheat bread; Rye + equal doses of inulin & gluten; Rye + low dose inulin + high dose gluten; Small non-supplemented rye
Other: Rye + equal doses of inulin & gluten — In a randomized cross-over design each subject receive one of six iso-caloric breakfasts on six different occasions, separated by 1 w wash-out.
  Arms: Large non-supplemented rye; Refined wheat bread; Rye + high dose inulin + low dose gluten; Rye + low dose inulin + high dose gluten; Small non-supplemented rye
Other: Rye + low dose inulin + high dose gluten — In a randomized cross-over design each subject receive one of six iso-caloric breakfasts on six different occasions, separated by 1 w wash-out.
  Arms: Large non-supplemented rye; Refined wheat bread; Rye + equal doses of inulin & gluten; Rye + high dose inulin + low dose gluten; Small non-supplemented rye
Other: Large non-supplemented rye — In a randomized cross-over design each subject receive one of six iso-caloric breakfasts on six different occasions, separated by 1 w wash-out.
  Arms: Refined wheat bread; Rye + equal doses of inulin & gluten; Rye + high dose inulin + low dose gluten; Rye + low dose inulin + high dose gluten; Small non-supplemented rye
Other: Small non-supplemented rye — In a randomized cross-over design each subject receive one of six iso-caloric breakfasts on six different occasions, separated by 1 w wash-out.
  Arms: Large non-supplemented rye; Refined wheat bread; Rye + equal doses of inulin & gluten; Rye + high dose inulin + low dose gluten; Rye + low dose inulin + high dose gluten
Other: Refined wheat bread — In a randomized cross-over design each subject receive one of six iso-caloric breakfasts on six different occasions, separated by 1 w wash-out.
  Arms: Large non-supplemented rye; Rye + equal doses of inulin & gluten; Rye + high dose inulin + low dose gluten; Rye + low dose inulin + high dose gluten; Small non-supplemented rye

SUMMARY:
Acute effects on appetite and metabolic function have been observed for whole-grain rye cereal products. The aim of this study is to evaluate if the appetite suppressing effect of a whole-grain rye breakfast cereal may be further enhanced by the addition of fermentable dietary fibre and plant protein. The aim is also to try to elucidate how observed effects on subjective appetite are mediated in terms of changes in hormonal signals, flow of nutrients in the blood and products from bacterial fermentation of dietary fibre, and to relate this to the different composition of the breakfasts.

DETAILED DESCRIPTION:
The short-term effects (up to 8 hours after intake) of dietary fibre and plant protein on subjective appetite and metabolism will be evaluated using a randomized cross-over study design. Each participant will consume six different breakfasts on six different occasions separated by a 1 week wash-out period: three rye porridges supplemented with three different combinations of added fermentable dietary fibre and plant protein, two non-supplemented rye porridges differing in amount of rye and one wheat bread. Participants will rate subjective appetite (satiety, hunger and desire to eat) by using a visual analog scale (VAS) every 30 min during an 8-hour period, starting 30 min before breakfast. The concentration of hydrogen and methane in the breath, as indicators of bacterial fermentation of dietary fibre, will be measured every hour. Blood samples will be collected before breakfast and at regular intervals throughout the day for analysis of glucose and hormone levels. The metabolic profile in the blood will be assessed as well as products from bacterial fermentation of dietary fibre, such as short chain fatty acids. Gastric emptying rate will also be evaluated using paracetamol as an indicator. Hormonal responses, changes in the metabolome and fermentation products will be related to subjective appetite and to differences in composition of the breakfasts.

ELIGIBILITY:
Inclusion Criteria:

* Women must be post-menopausal or habitually take hormonal contraceptives
* Habitual breakfast eaters

Exclusion Criteria:

* Non-contraceptive use among pre-menopausal women
* Pregnancy, lactation or wishing to become pregnant during the study period
* Dieting
* Weightloss
* Eating disorder
* Hyperglycemic
* Hyperinsulinemic
* Thyroid disease
* Metabolic issues
* Diabetes
* Physical or psychological problems eating
* Food intolerances/allergies to foods included in the study
* Vegetarians
* Intolerance/allergy to paracetamol
* Heavy smokers
* Recent or concurrent participation in an intervention research study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2013-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Subjective appetite profiles | 8 h (-30, 0, 30, 60, 90, 120, 150, 180, 210, 240, 270, 300, 330, 360, 390, 420, 450, 480)
  Subjective feelings of appetite (satiety, hunger and desire to eat) are assessed by visual analogue scale (VAS) (in total 18 measurements).

SECONDARY OUTCOMES:
Breath hydrogen and methane response | 8 h (-30, 30, 90, 150, 210, 270, 330, 390, 450, 480)
  Measurements of the concentration of breath hydrogen and methane(in total 10 measurements).
Gastric emptying rate | 8 h (-15, 15, 35, 65, 95, 125, 185, 230, 275, 305, 365, 470)
  Paracetamol (1 g) was taken with breakfast. The appearance of paracetamol in the blood is directly related to the rate of gastric emptying.
Glucose and hormonal response | 8 h (-15, 15, 35, 65, 95, 125, 185, 230, 275, 305, 365, 470)
  Glucose, insulin, glucagon, glucagon-like peptide-1 (GLP-1), glucose-dependent insulino-tropic polypeptide (GIP), peptide YY (PYY), cholecystokinin (CCK), leptin and ghrelin are measured in plasma samples.
Metabolic profiles | 8 h (-15, 15, 35, 65, 95, 125, 185, 230, 275, 305, 365, 470)
  The flux of nutrients is measured in plasma samples.
Products from bacterial fermentation of dietary fibre | 8 h (-15, 15, 35, 65, 95, 125, 185, 230, 275, 305, 365, 470)
  Products from bacterial fermentation of dietary fibre are measured in plasma samples.
Ad libitum food intake | 8 h after breakfast (480 min)
  Energy intakes will be assessed from the ad libitum dinner in order to validate subjective appetite measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Rikard K Landberg, Ass. Prof., Principal Investigator — Swedish University of Agricultural Sciences
Locations (1):
- Paediatric Research Facility; The Children's Hospital at Uppsala University Hospital, Uppsala, Uppsala County, Sweden